CLINICAL TRIAL: NCT04467775
Title: Sagittal Balance Through Ages
Acronym: ESTA
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7624
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2020-07

CONDITIONS: Spinal Deformity
Keywords: Spinal Deformity; Low back pain; Sciatica; Cervico brachial neuralgia
MeSH Terms: conditions — Low Back Pain; Sciatica; Brachial Plexus Neuritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The parameters of the sagittal balance of the cervical, thoracic and lumbar spine vary according to the types of spino-pelvic organization (types 1-4 according to Roussouly). These parameters have been described as a function of age in previous scientific work without taking into account the pelvic anatomy (pelvic incidence and spino-pelvic organization). This work, carried out within the framework of a round table of the French Society of Spinal Surgery (SFCR), would make it possible to provide a more detailed repository of existing radiographic parameters.

ELIGIBILITY:
Inclusion criteria:

* Minor or major subject aged 5 to 100
* Subject having carried out a telecolonne or EOS type X-ray for spinal balance (low back pain, sciatica, cervico-brachial neuralgia, inequality of length of the lower limbs) in spinal surgery consultation
* Subject not having expressed its opposition, after information, to the re-use of its data for the purposes of this research.

Exclusion criteria:

* Subject with surgical history, fractures, osteoporotic packing, vertebral deformation (scoliosis, kyphosis, spondylolisthesis grades 2-5), vertebral osteolysis (spondylodiscitis, tumor or metastasis).
* Subject who expressed his opposition to participate in the study
* Subject under guardianship or curatorship
* Subject under judicial protection

Ages: 5 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subject having carried out a telecolonne or EOS type X-ray for spinal balance (low back pain, sciatica, cervico-brachial neuralgia, inequality of length of the lower limbs) in spinal surgery consultation
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Retrospective study of the radiographic parameters measured by the KEOPS software | files analysed retrospectily from from January 1, 2014 to December 31, 2019 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie du Rachis, Strasbourg, France

REFERENCES:
- [Derived] Charles YP, Prost S, Pesenti S, Ilharreborde B, Bauduin E, Laouissat F, Riouallon G, Wolff S, Challier V, Obeid I, Boissiere L, Ferrero E, Solla F, Le Huec JC, Bourret S, Faddoul J, Abi Lahoud GN, Fiere V, Vande Kerckhove M, Campana M, Lebhar J, Giorgi H, Faure A, Sauleau EA, Blondel B; French Spine Surgery Society (SFCR). Variation of cervical sagittal alignment parameters according to gender, pelvic incidence and age. Eur Spine J. 2022 May;31(5):1228-1240. doi: 10.1007/s00586-021-07102-w. Epub 2022 Jan 6. PMID 34989876